CLINICAL TRIAL: NCT06911697
Title: In Vivo Detection of c-Met Activation Status by Specific PET/CT Imaging Based on 18F Labeled Small Molecule TKI
Brief Title: Study on c-Met Targeted PET/CT Imaging in NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xilin Sun (Other)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xilin Sun, Director, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-LLSC-23; 2023-LLSC-23 (Other: HarbinMU)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: PET/CT Imaging; NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: 18F-TSPF (Experimental): Each subject receives interval imaging of 18F-TSPF PET/CT and 18F-FDG PET/CT.
  Interventions: Diagnostic Test: 18F-TSPF PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-TSPF PET/CT — Each subject receives interval imaging of 18F-TSPF PET/CT and 18F-FDG PET/CT, and further follow-up.

SUMMARY:
The investigators developed a 18F labeled small molecule, 18F-TSPF, based on c-Met TKI, as a targeted molecular imaging agent for noninvasive and repeatable detecting c-Met activation status.

DETAILED DESCRIPTION:
In the study, NSCLC patients with different c-Met activation status (c-Met overexpression, MET exon 14 skipping mutation, MET amplification, MET wild type) confirmed by pathology or gene detection will receive 18F-TSPF PET/CT and 18F-FDG PET/CT respectively. The goal of the study is to evaluate specificity and accuracy of 18F-TSPF as a novel PET radiotracer to detect c-Met activation status and potentially identify c-Met-TKIs benefited NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years, open to both male and female participants;
2. Normal hepatic/renal function and cardiac function;
3. Expected survival of at least 12 weeks;
4. Good adherence to follow-up;
5. Presence of at least one measurable target lesion according to RECIST 1.1 criteria;
6. Women of childbearing age (15-49 years) must undergo a pregnancy test within seven days prior to the commencement of the study and test negative; sexually active male and female participants must agree to utilize effective contraception to prevent pregnancy during the study and for three months following the final examination;
7. Patients for whom a clinical physician recommends PET/CT scans for the diagnosis and staging of tumors;
8. Participants must fully understand and voluntarily agree to participate in the study, and must sign an informed consent form.

Exclusion Criteria:

1. Severe abnormalities in liver and renal function and blood counts;
2. Patients planning to conceive;
3. Pregnant or lactating women;
4. Individuals unable to lie flat for thirty minutes;
5. Individuals who refuse to participate in this clinical study;
6. Individuals suffering from claustrophobia or other psychiatric disorders;
7. Other situations deemed unsuitable for trial participation by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Values | 1 hour
  To quantify the PET, a volume of interest using a 3-D sphere, was placed over the primary lung tumor, lymph nodes and distant metastases avoiding necrosis, blood vessels and normal lung tissue as much as possible on a workstation (Advantage Workstation 4.6; GE Healthcare). The maximum standard uptake value (SUVmax) normalized to body weight (kBq/mL) was calculated within the region of interest. SUVmax of primary lesion and metastatic lesion in subjects with NSCLC are measured and used to analyze correlatation with pathology or gene detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Yes
Xilin Sun
Supporting Information: Study Protocol